CLINICAL TRIAL: NCT04755803
Title: A Prospective Registry of Patients With Congenital Penile Anomalies
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kwanjin Park, Principal Investigator, Seoul National University Hospital
Other Study IDs: 2008-057-1147
Record Dates: First submitted 2021-02-09; First posted 2021-02-16 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Concealed Penis; Hypospadias; Phimosis; Chordee
MeSH Terms: conditions — Hypospadias; Phimosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Dartos Fascia is commonly known as subcutaneous tissue of the penis. It is located under the foreskin and superficially located on the outer external spermatic fascia of the scrotum and the axis of the penis. The primary role of dartos fascia is the mobility of the foreskin in the basal tissue and the blood supply from the external sinus vessels. Furthermore, it promotes heat loss and cools down the testicles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Penoplasty — Modified penoplasty technique:
  1. Degloved the penile skin and excise the inner prepuce.
  2. Advanced penoscrotal skin to cover penile shaft
  3. Fixed the penis base and reconstructed the penoscrotal angle

SUMMARY:
Prospective registry and biobank in pediatric patients with congenital penile anomalies

DETAILED DESCRIPTION:
According to the U.S. Center for Disease Control and Prevention, in the United States, one in 200 babies is born with congenital penile anomalies. In Korea, there is a rapid increase rate among other types of congenital anomalies from 1993 to 2010, from 0.7 to 10,000 to 9.9 per 10,000 cases. It leaves long term sequelae into adulthood even after the corrective operation has been performed. Some of the sequelae that patients experienced were difficulties in micturition, dissatisfaction with the appearance of the penis, and decreased sexual function, as well as psychosexual well-being.

Despite its high prevalence, hypospadias and related penile anomalies have no specific known etiology and mechanisms. However, numerous studies have shown that both gene and environment play a significant role in making etiologies multifactorial. Furthermore, a molecular trial shows that both genetics and environmental factors disrupt the normal development course of the phallus, or penis. Penis formation, growth, or the formation of the male urogenital system, in general, have shown to be androgen dependent. Any defect in the androgen synthesis leading to androgen deficiency or receptors may play a role, specifically, in the development of penile anomalies.

Pediatric patients between the ages of 0 to 18 years, with congenital penile anomalies and scheduled to undergo penoplasty will be enrolled. In this prospective observational study, our aims are to collect dartos fascia, which is a tissue in penile region, and examine histochemistry of the sample.

ELIGIBILITY:
Inclusion Criteria:

* Those with congenital penile anomalies (e.g. hypospadias, chordee, webbed penis) and receiving penoplasty at the institution.
* Those who understand the registry's content and are signed and dated by the patient (or the patient's legal guardian or representative).

Exclusion Criteria:

* Those who are unwilling to participate and do not sign the informed consent.
* Unable to read or understand Korean.

Ages: 0 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This registry is gender-specific and only males with congenital penile anomalies and receiving penoplasty at the institution are allowed to be enrolled.
Study Population: Male patients between the ages of 0 to 18 years with congenital penile anomalies and receiving penoplasty at the institution.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Dartos Fascia (Penile Tissue) sample collection | Procedure (At the time of penoplasty)
  Collection of biological samples from pediatric patients who have been registered onto the prospective registry.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No